CLINICAL TRIAL: NCT01403129
Title: Early Detection of Keratoconus Using Ultrasound
Brief Title: Keratoconus Detection by Ultrasound
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ronald H Silverman, Professor of Ophthalmic Science, Columbia University
Other Study IDs: AAAF1497; R01EY019055 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Keratoconus
Keywords: keratoconus; keratoconus-suspect; ultrasound exam; acoustic radiation force ultrasound exam
MeSH Terms: conditions — Keratoconus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Keratoconus-Suspect: A person who has or is suspected of having keratoconus. Will have either or both Artemis-2 exam and OCT exam.
  Interventions: Procedure: Artemis Ultrasound Exam; Procedure: Optical Coherence Tomography (OCT) Exam
- Keratoconus-Related: A person who is genetically related to someone with keratoconus. Will have either or both Artemis-2 exam and OCT exam.
  Interventions: Procedure: Artemis Ultrasound Exam; Procedure: Optical Coherence Tomography (OCT) Exam
- Age-Matched Normal: A person who is approximately the same age as subjects who have been enrolled in the study.
  Will have either or both Artemis-2 exam and OCT exam.
  Interventions: Procedure: Artemis Ultrasound Exam; Procedure: Optical Coherence Tomography (OCT) Exam

INTERVENTIONS:
Procedure: Artemis Ultrasound Exam — Ultrasound exam of both eyes using an Artemis-2 device. Exam will be performed once. Exam duration is 20 minutes per eye.
  Other Names: Ultrasound biomicroscope (UBM); High frequency ultrasound
Procedure: Optical Coherence Tomography (OCT) Exam — OCT exam of both eyes. Exam will be performed once, duration is 10. I utes per eye.
  Other Names: OCT

SUMMARY:
Keratoconus (KC) is a corneal disease which will in many cases ultimately require corneal transplantation to maintain vision. Early detection, which is not possible with current technology, would allow early treatment and prevent severe damage to KC corneas inadvertently operated upon for correction of vision. The investigators' aim is to combine measurements of different properties of the cornea to develop means for early detection of KC.

DETAILED DESCRIPTION:
Keratoconus is the most common degenerative disease affecting the cornea. As keratoconus develops, the cornea thins and bulges. Eventually, a corneal transplant may be needed to maintain vision. In its earliest stages, the disease is particularly difficult to detect. This is of great importance to the corneal refractive surgeon because surgical treatment of a keratoconic cornea will weaken it and greatly accelerate the occurrence of symptoms. Early detection of keratoconus will benefit patients because of the recent development of methods for strengthening the corneal stroma and preventing disease progression.

The investigators have developed a technique based on the use of high resolution ultrasound for imaging the cornea and measuring the thickness of its component layers, including the epithelium and the stroma. In early keratoconus, as the anterior stromal surface begins to bulge forward, the epithelium will thin above the apex of the bulge and thicken around it, to maintain a smooth anterior surface. The investigators have also developed methods for characterizing the elastic properties of the cornea by inducing and measuring surface displacements in response to a pulse of acoustic radiation force.

The investigators' goal is to reduce the percentage of screened cases deemed keratoconus-suspect by at least a factor of two by allowing an unambiguous diagnosis of early keratoconus. This would provide two major benefits; (1) to be able to predict eyes with higher risk of developing ectasia after corneal refractive surgery, and (2) early diagnosis would allow earlier treatment of the condition with collagen crosslinking, preserving the cornea from disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of keratoconus (KC) or keratoconus-suspect
* Blood relation of person with KC
* Age-matched normal of KC subjects
* Ability to sit still in front of ultrasound unit and lie on exam table

Exclusion Criteria:

* Other eye disease

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to CUMC associated physicians and the London Vision Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-12; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Differences in elastic parameters between normal and KC corneas. | Up to 1 year after enrollment
  The undamped vibrational frequency and damping time-constant for the anterior and posterior corneal surfaces and for Bowman's membrane will be measured. The elastic modulus will be calculated form the change in corneal thickness resulting from known radiation force.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Silverman, PhD, Principal Investigator — Columbia University
Locations (2):
- Columbia University Medical Center, New York, New York, United States
- London Vision Clinic, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Urs R, Lloyd HO, Silverman RH. Acoustic radiation force for noninvasive evaluation of corneal biomechanical changes induced by cross-linking therapy. J Ultrasound Med. 2014 Aug;33(8):1417-26. doi: 10.7863/ultra.33.8.1417. PMID 25063407
- [Result] Silverman RH, Urs R, Roychoudhury A, Archer TJ, Gobbe M, Reinstein DZ. Epithelial remodeling as basis for machine-based identification of keratoconus. Invest Ophthalmol Vis Sci. 2014 Mar 13;55(3):1580-7. doi: 10.1167/iovs.13-12578. PMID 24557351
- [Result] Ursea R, Feng M, Urs R, RoyChoudhury A, Silverman RH. Comparison of artemis 2 ultrasound and Visante optical coherence tomography corneal thickness profiles. J Refract Surg. 2013 Jan;29(1):36-41. doi: 10.3928/1081597X-20121126-01. Epub 2012 Nov 30. PMID 23205905
- [Result] Urs R, Lloyd HO, Reinstein DZ, Silverman RH. Comparison of very-high-frequency ultrasound and spectral-domain optical coherence tomography corneal and epithelial thickness maps. J Cataract Refract Surg. 2016 Jan;42(1):95-101. doi: 10.1016/j.jcrs.2015.07.038. PMID 26948783
- [Result] Reinstein DZ, Archer TJ, Urs R, Gobbe M, RoyChoudhury A, Silverman RH. Detection of Keratoconus in Clinically and Algorithmically Topographically Normal Fellow Eyes Using Epithelial Thickness Analysis. J Refract Surg. 2015 Nov;31(11):736-44. doi: 10.3928/1081597X-20151021-02. PMID 26544561
- [Result] Reinstein DZ, Yap TE, Archer TJ, Gobbe M, Silverman RH. Comparison of Corneal Epithelial Thickness Measurement Between Fourier-Domain OCT and Very High-Frequency Digital Ultrasound. J Refract Surg. 2015 Jul;31(7):438-45. doi: 10.3928/1081597X-20150623-01. PMID 26186562
- [Result] Silverman RH, Urs R, RoyChoudhury A, Archer TJ, Gobbe M, Reinstein DZ. Combined tomography and epithelial thickness mapping for diagnosis of keratoconus. Eur J Ophthalmol. 2017 Mar 10;27(2):129-134. doi: 10.5301/ejo.5000850. Epub 2016 Aug 8. PMID 27515569
- See also: Ronald H. Silverman Homepage — http://columbiaeye.org/profile/rhsilverman?profile=researcher
- See also: Dan Z. Reinstein Homepage — http://www.londonvisionclinic.com/blog/dan-reinstein/